CLINICAL TRIAL: NCT06388616
Title: A Phase I, Single-Dose, Non-Randomised, Open-Label, Parallel-Group Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics, Safety, and Tolerability of Balcinrenone
Brief Title: Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics, Safety, and Tolerability of Balcinrenone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6402C00013
Record Dates: First submitted 2024-04-16; First posted 2024-04-29 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; Healthy participants; Balcinrenone; Pharmacokinetics; Safety
MeSH Terms: interventions — AZD9977

STUDY DESIGN:
Intervention Model Description: Three cohorts (two hepatic impairment cohorts and controls with normal hepatic function) will be enrolled into this study.
  All subjects will receive the study intervention:
  * Cohort 1 will enroll 8 participants with mild hepatic impairment
  * Cohort 2 will enroll 8 participants with moderate hepatic impairment
  * Cohort 3 will enroll 8-12 healthy participants matched on a group level regarding age, BMI and sex
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Subjects with Mild Impairment will receive a single oral dose of balcinrenone under fasted conditions.
  Interventions: Drug: Balcinrenone
- Group 2 (Experimental): Subjects with Moderate Impairment will receive a single oral dose of balcinrenone under fasted conditions.
  Interventions: Drug: Balcinrenone
- Group 3 (Experimental): Healthy participants will receive a single oral dose of balcinrenone under fasted conditions.
  Interventions: Drug: Balcinrenone

INTERVENTIONS:
Drug: Balcinrenone — 50 mg, Immediate release capsule to be taken orally.
  Other Names: AZD9977

SUMMARY:
This study will evaluate the pharmacokinetics (PK), safety, and tolerability of a single oral dose of balcinrenone in patients with mild and moderate hepatic impairment in comparison to a matched healthy control group.

DETAILED DESCRIPTION:
This is an open-label, non-randomised, multicentre, parallel-group, single-dose study to examine the PK, safety, and tolerability of balcinrenone 50 mg administered orally to male and female participants with mild or moderate hepatic impairment compared with control participants with normal hepatic function. Eight participants with mild impairment and 8 participants with moderate impairment per CP classification and 8 to 12 participants with normal hepatic function matched on a group level regarding age, BMI, and sex to the impaired groups are planned for study intervention. All participants will receive a single dose of balcinrenone 50 mg on Day 1 following an overnight fast. Study intervention will be administered orally with approximately 240 mL of water.

Child-Pugh scoring will be used to determine the level of hepatic impairment. Participants will be enrolled into the following groups based on their CP classification score as determined at screening:

* Group 1: Participants with mild hepatic impairment (CP Class A, score of 5 or 6).
* Group 2: Participants with moderate hepatic impairment (CP Class B, score of 7 to 9).
* Group 3: Participants with normal hepatic function matched on a group level regarding age, BMI, and sex to the impaired groups.

ELIGIBILITY:
Inclusion Criteria:

- Participant must be 18 to 79 years of age, inclusive, at the time of signing the informed consent.

For participant with hepatic impairment:

* Participant must have a diagnosis of chronic (≥ 6 months) and stable hepatic impairment Child Pugh Class A or B (eg, no clinically significant change in signs, symptoms, or laboratory parameters of hepatic disease status within 30 days prior to study screening, as determined by the investigator at screening and Day -1).
* Supporting documents confirming the participant's hepatic impairment must be available; participant self-report is not acceptable; the participant must be classified by the investigator as CP Class A or B at screening.
* Participants must be stable on a concomitant medication and/or treatment regimen (defined as not starting a new treatment/medication[s] or a change in the dosage or frequency of the concomitant medication[s] within 2 weeks prior to screening). Minor changes in dosage can be accepted at the discretion of the investigator.

For participant with normal hepatic function:

* Participant must be medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or 12-lead ECGs, as deemed by the investigator at screening and Day -1.
* Body weight ≥ 50 kg; BMI within the range of 18.0 to 42.0 kg/m2 (inclusive) as measured at screening.
* Sex: male and female.
* Females must not be lactating and must not have a positive pregnancy test at screening and at Day -1.
* Women of childbearing potential (defined as female participants who are neither permanently sterilised [hysterectomy, bilateral oophorectomy, or bilateral salpingectomy] nor postmenopausal) must use a highly effective method of contraception (described below).
* A highly effective method of contraception is defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly. Women of childbearing potential who are sexually active with a non-sterilised male partner must agree to use one highly effective method of birth control, as defined below, from enrolment throughout the study and until at least 4 weeks after study intervention.
* Highly effective methods of contraception include: sexual abstinence (periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods], declaration of abstinence for the duration of exposure to IMP, and withdrawal [coitus interruptus], spermicides only, and lactational amenorrhoea method are not acceptable methods of contraception), a vasectomised partner, bilateral tubal occlusion, combined (oestrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device, intrauterine hormone-releasing system.
* Women of nonchildbearing potential (defined as female participants who are permanently surgically sterilised [hysterectomy, bilateral oophorectomy, or bilateral salpingectomy] or postmenopausal).
* Women will be considered postmenopausal if they have been amenorrhoeic for 12 months prior to the planned date of study intervention without an alternative medical cause. The following age-specific requirements apply:
* Women < 55 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatment and FSH levels in the postmenopausal range.
* Women ≥ 55 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatment.
* Postmenopausal status for participants with hepatic impairment based on FSH levels may be at the discretion of the investigator.
* Capable of giving signed informed consent as described in Appendix A which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
* Provision of signed and dated written ICF prior to any mandatory study-specific procedures, sampling, and analyses.

Exclusion Criteria:

* Participant has eGFR < 60 mL/minute/1.73 m2 as calculated by CKD-EPI.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the investigator at screening or Day -1, or history of hypersensitivity to drugs with a similar chemical structure or class to balcinrenone.
* History of long QT syndrome or any clinically significant abnormalities on 12-lead ECG at screening or Day -1, as judged by the investigator, including but not limited to any of the following:
* Any significant arrhythmia.
* Conduction abnormalities (eg, Wolff Parkinson White syndrome, second degree AV block; at the discretion of the investigator).
* Prolonged QTcF > 450 ms for participants with normal hepatic function; > 480 ms for participants with mild or moderate hepatic impairment.
* Clinically significant PR (PQ) interval shortening (< 120 ms) or prolongation (> 240 ms); intermittent second or third degree AV block, or AV dissociation.
* Complete bundle branch block and/or QRS duration > 120 ms.
* Any of the following signs or confirmation of COVID-19 infection at screening or Day -1:
* Participant has a positive SARS-CoV-2 test result within 2 weeks prior to screening, at screening, or on Day -1.
* Clinical signs and symptoms consistent with COVID-19 (eg, fever, dry cough, dyspnoea, sore throat, fatigue) within 2 weeks prior to screening or Day -1.
* Positive test for HIV at screening.
* Positive results at screening for hepatitis B surface antigen, hepatitis B core antibody or hepatitis C virus. Participants with impaired hepatic function with positive total hepatitis B core antibody or positive hepatitis C result may be included if a follow-up hepatitis B virus DNA test or follow-up hepatitis C virus RNA test is negative.
* History or presence of clinically significant thyroid disease, in the opinion of the investigator. Participants with clinically significant TSH levels outside normal limits at screening will not be enrolled. Participants on stable thyroid replacement therapy are not excluded.
* History or presence of clinically significant or unstable medical or psychiatric condition or disease in the opinion of the investigator.
* Participant is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or Day -1 or expected during the conduct of the study.
* History of any major surgical procedure within 30 days prior to study intervention.
* Any clinically or surgically significant condition that may affect balcinrenone absorption and/or excretion in the opinion of the investigator, including gastric restrictions and bariatric surgery (eg, gastric bypass). Uncomplicated appendectomy and hernia repair will be allowed. Uncomplicated cholecystectomy is allowed at the discretion of the investigator.
* Judgment by the investigator that the participant should not participate in the study if they have any ongoing or recent (ie, during the screening period) minor medical complaints that may interfere with the interpretation of study data or if they are considered unlikely to comply with study procedures, restrictions, and requirements.
* Use of any medication defined as prohibited medication (see Appendix E) within 2 weeks prior to study intervention or longer if the medication has a long half-life.
* Unable to refrain from the following for 10 hours prior to and 10 hours after study intervention: Phosphate binders (eg, aluminium hydroxide and calcium carbonanate).

Acid reducing agents (eg, ranitidine/nizatidine or proton pump inhibitors). Cholestyramine/colestipol. MRA agents (eg, spironolactone, eplerenone, finerenone).

* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days of study intervention in this study or, if known, 5 half-lives from last dose in the previous study to study intervention in this study, whichever is longest.
* Previous enrolment in the present study. Note: participants consented and screened, but not receiving study intervention in this study or a previous Phase I study, are not excluded.
* Participant smokes more than 10 cigarettes (ie, 1/2 pack) per day or equivalent (eg, e-vapor cigarette, pipe, cigar, chewing tobacco, nicotine patch, nicotine gum) and is unable to comply with the nicotine restrictions (Section 5.3.2) during the study.
* Positive screen for drugs of abuse (unless participant has hepatic impairment and positive screen is due to medication[s] prescribed by physician) and/or alcohol test at screening or Day -1.
* Receipt of blood products within 2 months prior to Day -1, plasma or platelets donation within 1 month prior to Day -1, or any blood donation/blood loss > 500 mL within 3 months prior to Day -1.
* Involvement of any AstraZeneca or clinical unit employee or their close relatives.
* Vulnerable participants, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
* Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.

Participants with hepatic impairment are excluded from the study if any of the following criteria apply:

* Esophageal banding within 3 months prior to Day -1 or required treatment for gastrointestinal bleeding within 6 months prior to Day -1.
* Ascites requiring paracentesis and albumin infusion at 4-week intervals or less.
* History of paracentesis within 30 days prior to screening.
* Fluctuating or rapidly deteriorating hepatic function, as indicated by strongly varying or worsening of clinical and/or laboratory signs of hepatic impairment within the screening period.
* In the opinion of the investigator, any evidence of additional severe or uncontrolled systemic disease (eg, currently unstable or uncompensated renal, cardiovascular, or respiratory disease) or laboratory finding that makes it unsafe for the participant to participate in the study.
* Presence of a hepatocellular carcinoma or acute liver disease caused by an infection or drug toxicity.
* Hepatic impairment due to non-liver disease (eg, right HF).
* Biliary obstruction or other causes of hepatic impairment not related to parenchymal disorder and/or disease of the liver.
* Clinically relevant hepatic encephalopathy (Grade 2 or more) at screening or Day -1.
* Has required new medication for hepatic encephalopathy within the 3 months prior to Day -1.
* Platelet count < 35 × 109/L and/or neutrophil count < 1.2 × 109/L and/or haemoglobin < 85 g/L.
* Current functioning organ transplant or anticipated to receive organ transplant within 2 months of screening or Day -1.
* Participant has had a porto-systemic shunt (including transjugular intrahepatic portosystemic shunts).
* History of drug abuse within 1 year prior to screening.
* History of alcohol abuse within 3 months prior to screening and/or consumes > 21 units per week for males and > 14 units per week for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.
* Supine systolic BP > 160 or <90 mmHg, and diastolic BP > 95 or < 40 mmHg at screening or Day -1. One repeat is allowed.
* Supine pulse rate < 50 bpm or > 99 bpm at screening or Day -1. One repeat is allowed.
* Cardiac bradyarrhythmia or tachyarrhythmia requiring treatment (atrial fibrillation/flutter with optimal control of ventricular rate is not excluded) at screening or Day -1.
* Blood dyscrasias with increased risk of bleeding including idiopathic thrombocytopenic purpura and thrombotic thrombocytopenic purpura or symptoms of increased risk of bleeding (frequent bleeding gums or nose bleeds) at screening or Day -1.
* History of unstable diabetes mellitus as evidenced by hemoglobin A1c ≥ 9% at screening.

Participants with normal hepatic function are excluded from the study if any of the following criteria apply:

* History of any clinically important disease or disorder, which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of dose administration.
* Any laboratory values with the following deviations at screening or Day -1

  (1 confirmatory repeat is allowed):
* ALT and/or AST > 1.2 × ULN.
* White blood cell count and/or platelet count < lower limit of normal; haemoglobin < 11.0 g/dL for females or < 12.0 g/dL for males.
* Activated partial thrombin time and prothrombin time (or INR) > 1.2 × ULN.
* Bilirubin > 1.5 × ULN (or known Gilbert's syndrome).
* Changes in any current medication (initiation, dose change, or cessation), that may impact the study readouts (as judged by the investigator) within 2 weeks prior to screening and until study intervention. This criterion does not apply to medication prescribed for occasional use.
* History or presence of hepatic disease or evidence of other known forms of known chronic liver disease, eg, alcoholic liver disease, hepatitis B, hepatitis C, primary biliary cirrhosis, primary sclerotic cirrhosis, autoimmune hepatitis, Wilson disease, iron overload, alpha-1-antitrypsin deficiency, drug-induced liver injury, known or suspected hepatocellular carcinoma.
* History of drug abuse within 2 years prior to screening.
* History of alcohol abuse within 2 years prior to screening and/or consumes > 21 units per week for males and > 14 units per week for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.
* Supine systolic BP > 150 or < 90 mmHg, and diastolic BP > 95 or < 50 mmHg at screening or Day -1. One repeat is allowed.
* Supine pulse rate < 45 bpm or > 100 bpm at screening or Day -1. One repeat is allowed.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from time zero to the last measurable concentration (AUClast) | Day 1 to Day 5
  To compare the PK of a single oral dose of balcinrenone in participants with mild and moderate hepatic impairment to those with normal hepatic function
Area under plasma concentration-time curve from zero to infinity (AUCinf) | Day 1 to Day 5
  To compare the PK of a single oral dose of balcinrenone in participants with mild and moderate hepatic impairment to those with normal hepatic function
Maximum observed plasma concentration (Cmax) | Day 1 to Day 5
  To compare the PK of a single oral dose of balcinrenone in participants with mild and moderate hepatic impairment to those with normal hepatic function

SECONDARY OUTCOMES:
AEs and SAEs up to the follow-up telephone call (Day 10 [± 3 days]) | Screening (day -28 to day -2) to day 10
  To assess the safety and tolerability of a single oral dose of balcinrenone in participants with mild and moderate hepatic impairment and those with normal hepatic function
Number of participants with abnormal Vital signs, abnormal ECGs, and abnormal physical examination findings | Screening (day -28 to day -2) to day 4
  To assess the safety and tolerability of a single oral dose of balcinrenone in participants with mild and moderate hepatic impairment and those with normal hepatic function
Number of participants with abnormal laboratory tests results | Screening (day -28 to day -2) to day 4
  To assess the safety and tolerability of a single oral dose of balcinrenone in participants with mild and moderate hepatic impairment and those with normal hepatic function

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Marbury, M.D., Principal Investigator — Servico Integrado de Tecnicas Endovasculares; Eric J Lawitz, M.D., Principal Investigator — Servico Integrado de Tecnicas Endovasculares; Juan C Rondon, M.D., Principal Investigator — Servico Integrado de Tecnicas Endovasculares
Locations (3):
- United States (3):
  - Research Site, Hialeah, Florida
  - Research Site, Orlando, Florida
  - Research Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home